CLINICAL TRIAL: NCT02345798
Title: Preparing Patients and Informal Caregivers for Lung Surgery: Pilot Study of a Video-Assisted Intervention to Enhance Post-Operative Recovery
Brief Title: Video-Assisted Intervention in Improving Recovery in Patients With Cancer Undergoing Lung Surgery and Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14302; NCI-2014-02539 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14302 (Other: City of Hope Medical Center)
Record Dates: First submitted 2014-12-22; First posted 2015-01-26 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Malignant Lung Neoplasm
MeSH Terms: conditions — Lung Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (standard care) (Active Comparator): Patients and caregivers receive standard care during routine clinic visits.
  Interventions: Procedure: Standard Follow-Up Care; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (video-assisted intervention) (Experimental): Patients view Parts 1 and 2 of the video program, which focus on what to expect before surgery and after surgery in the hospital, on a tablet over approximately 8 minutes at a scheduled pre-operative visit. Patients then receive an educational handbook and discuss the video with a nurse. After surgery and before hospital discharge, patients view Part 3 of the video over approximately 6 minutes, which focuses on what to expect after going home.
  Interventions: Other: Caregiver-Related Intervention or Procedure; Other: Educational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Standard Follow-Up Care — Undergo usual care
  Arms: Arm I (standard care)
Other: Caregiver-Related Intervention or Procedure — Undergo video-assisted intervention
  Arms: Arm II (video-assisted intervention)
Other: Educational Intervention — Undergo video-assisted intervention
  Other Names: Education for Intervention; Intervention, Educational
  Arms: Arm II (video-assisted intervention)
Other: Quality-of-Life Assessment — Undergo quality of life assessment
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Undergo questionnaire administration

SUMMARY:
This pilot clinical trial studies a video-assisted intervention in improving recovery of patients undergoing surgery to remove lung cancer or cancer that has spread to the lung and their caregivers. The intervention uses educational videos to prepare patients and families for surgery and teach them how to manage the symptoms after surgery. Teaching patients and their families what to expect before and after surgery may help improve patient and caregiver quality of life, help patients recover better from surgery, and support families in their role as caregivers after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To pilot test a video-assisted intervention designed to enhance post-operative recovery by preparing patients and informal caregivers for lung surgery.

SECONDARY OBJECTIVES:

I. To describe preliminary effect of the video-assisted intervention on patient-reported outcomes (PROs), informal caregiver-reported outcomes, and clinical/system outcomes.

OUTLINE: Patients and their caregivers are assigned to 1 of 2 arms.

ARM I: Patients and caregivers receive standard care during routine clinic visits.

ARM II: Patients view Parts 1 and 2 of the video program, which focus on what to expect before surgery and after surgery in the hospital, on a tablet over approximately 8 minutes at a scheduled pre-operative visit. Patients then receive an educational handbook and discuss the video with a nurse. After surgery and before hospital discharge, patients view Part 3 of the video over approximately 6 minutes, which focuses on what to expect after going home.

After completion of study, patients and caregivers are followed up at approximately 2-4 weeks and 2 months.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS: Scheduled to undergo surgery with lung resection for treatment of primary or secondary neoplasms of the lung
* PATIENTS: Able to read and understand English
* INFORMAL CAREGIVERS: The primary informal caregiver as identified by patients participating in the study; this refers to either a family member or friend who will be providing the majority of care following surgery
* INFORMAL CAREGIVERS: Able to read and understand English
* This protocol is eligible for waiver of informed consent documentation; all subjects must have the ability to understand and the willingness to provide verbal informed consent

Exclusion Criteria:

* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
Patient-reported outcomes to video-assisted intervention among the lung surgery population at City of Hope (COH) | Up to 2 months
  Patient-reported outcomes assessed using the State Trait Anxiety Inventory (STAI), For all patient-reported outcomes, data will be summarized using descriptive statistics of mean and standard deviation.
Informal caregiver-reported outcomes to video-assisted intervention among the lung surgery population at COH | Up to 2 months
  Informal caregiver-reported outcomes assessed using the STAI. For all informal caregiver-reported outcomes, data will be summarized using descriptive statistics of mean and standard deviation.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Kim, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States